CLINICAL TRIAL: NCT05023785
Title: The Harmonized Interventions to Maintain Health Via Appropriate Risk Factor Modification and Lifestyle Changes in Pediatric, Adolescent and Young Adult Cancer Survivors Study: A Multicentre Randomized Controlled Trial
Brief Title: The HIMALAYAS Trial and Lifestyle Changes in Pediatric, Adolescent and Young Adult Cancer Survivors Study: A Multicentre Randomized Controlled Trial
Acronym: HIMALAYAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Centre hospitalier de l'Université de Montréal (CHUM) (Other); Queen Elizabeth II Health Sciences Centre (Other); Alberta Health services (Other); Vancouver General Hospital (Other); Université de Montréal (Other); Dalhousie University (Other); University of Alberta (Other); University of British Columbia (Other); University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-5626
Record Dates: First submitted 2021-04-29; First posted 2021-08-27 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure; Cardiotoxicity; Cancer
Keywords: Adolescents and Young Adults; Exercise Therapy; Behavioral and Peer Support; Cardiac Rehabilitation; Cancer Survivor
MeSH Terms: conditions — Heart Failure; Cardiotoxicity; Neoplasms; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardio-Oncology Rehabilitation (CORE) (Experimental): Participants in the CORE group will have
  1. A personalized, supervised exercise program ((in-person at intuition and virtual/ homebased exercises)
  2. CV risk factor management,
  3. behavioural support for the first 6 months. The behavioural support will continue for CORE participants from months 7-24. Behavioural support includes professionally guided and peer-enhanced exercise behavioural support based on behaviour change stage theories.
  CORE participants will be provided a wrist-worn heart and physical activity monitor to use throughout the 24-month observation period.
  Interventions: Behavioral: Cardio-oncology Rehabilitation (CORE)
- Standard of Care (CON) (No Intervention): Participants in the CON group will receive standard medical care and physical activity will be monitored by a wrist-worn activity tracker for 2 years.

INTERVENTIONS:
Behavioral: Cardio-oncology Rehabilitation (CORE) — Exercise therapy, CVD risk factor management for the first 6 months (as per current standards in CR models) and behavioural support for the entire 2-year intervention period
  Arms: Cardio-Oncology Rehabilitation (CORE)

SUMMARY:
Pediatric, adolescent and young adult cancer survivors (PAYA-CS) are at higher risk of cardiovascular (CV) morbidity and mortality. This is a consequence of prior cancer-related therapies that have the potential of producing cardiac dysfunction, reducing cardiorespiratory fitness (reduced VO2peak) and psychosocial morbidities (i.e., anxiety and depression). A reduction of physical activity levels can evoke functional limitations resulting in a vicious cycle of reduced exercise tolerance and physical deterioration. To date, there is limited evidence on the use of non-pharmacological strategies such as Cardio-Oncology Rehabilitation (CORE) including structured exercise, behavioural support and risk factor management to improve the outcomes of this underserved population. The HIMALAYAS study is a randomized controlled trial designed to evaluate the impact of a CORE intervention (consisting of six-months home and onsite-based structured moderate to high-intensity aerobic exercise training and CVD risk factor management) on CV and psychosocial health, and the cardiovascular disease risk in PAYA-CS with mild heart dysfunction (stage B heart failure) compared to standard of care (i.e. providing guidance on the current exercise recommendations for cancer survivors). The primary objective of the HIMALAYAS study is to determine whether a six-month supervised CORE intervention, consisting of individualized moderate to high-intensity aerobic exercise training, CVD risk factor modification and enhanced online behavioral support, improves cardiorespiratory fitness (VO2peak; primary outcome), cardiac function, CVD risk factors and biomarkers, and patient-reported outcomes (PROs) at six- months follow-up compared to standard of care (CON) in PAYA-CS with stage B heart failure. The secondary objective is to assess the same outcomes at 12- and 24-months follow-up. We will recruit 336 patients across 5 sites in Canada and upto 134 patients at UHN in 3 years and conclude in 6 years.

DETAILED DESCRIPTION:
Over 90,000 North Americans are diagnosed with cancer before the age of 40. Improved cancer therapies have led to an exponential growth in the number of pediatric, adolescent, and young adult cancer survivors (AYA-CS) who are expected to live 50-60 years beyond diagnosis. However, AYA-CS are at increased risk of developing multiple cancer- and treatment-related morbidities including poor fitness (e.g., low VO2peak), hypertension (HTN), diabetes, and poor mental health, which all contribute to premature cardiovascular disease (CVD). The prevalence of CVD events (e.g. heart failure, heart attack, stroke) is up to 23.8% in adult survivors of pediatric cancers with long term follow-up after treatment. The incidence of subclinical CVD, which is a precursor to CVD events, is even higher in AYA-CS; up to 40%, 11%, and 5% experience subclinical cardiomyopathy measured by abnormal global longitudinal strain (GLS), diastolic dysfunction (DD) or mild reduction in left ventricular ejection fraction (LVEF), respectively, and 18% experience reduced aerobic fitness. The treatment of modifiable CVD risk factors must be considered a fundamental target for improving CVD health-related outcomes in AYA-CS. To this end, exercise and best-practices for CVD risk factor modification are integral to a cardiac rehabilitation model. Traditional cardiac rehabilitation models for patients with CVD (consisting of exercise, CVD risk factor treatment, and patient education) are safe and effective in improving HRQoL, morbidity, and mortality risk. However, by virtue of their age and low short-term CVD risk, AYA-CS do not meet traditional criteria for initiating cardiac rehabilitation (CR) and are less likely to receive treatments to reduce CVD risk. AYA-CS with stage B heart failure (SBHF): (1) are at high risk for subsequent HF/CVD death; (2) have lower cardiopulmonary fitness; and (3) are more likely to benefit from CVD risk factor management. Considering that AYA-CS have an estimated 33% prevalence of SBHF, this vulnerable cohort of cancer survivors represent an opportunity for intervention that is highly feasible and potentially impactful. Exercise is a preferred method for optimizing health and survival in PAYA-CS. However, we need models that safely and effectively deliver exercise interventions that meet the unique needs of this population. The cardio-oncology rehabilitation (CORE) model is an intervention that would provide AYA-CS with SBHF a supervised and home-based high-intensity interval training (HIIT) and moderate-intensity continuous training (MICT) exercise therapy, CVD risk factor modification, and behavioural support to reduce the risk of CVD. The primary objective of the HIMALAYAS study is to determine whether supervised CORE (Group 1A) improves cardiorespiratory fitness (VO2peak; primary outcome), cardiac function, CVD risk factors and biomarkers, and PROs at 6 months (primary timepoint) as well as 12 and 24 months compared to standard of care group control group (CON) in AYA-CS with SBHF.

The secondary objective of the study is to assess the ongoing behavioural support strategy based on the exercise guidelines for cancer survivors (i.e. 90 to 150 minutes of moderate to vigorous PA per week) on VO2peak, cardiac function, CVD risk factors and biomarkers, and PROs at 24 months compared to standard of care [CON] in AYA-CS with SBHF. Due to the COVID-19 pandemic, CORE intervention will involve a facility-based HIIT session and home-based HIIT session (described as "HIIT at Home") per week.

ELIGIBILITY:
Inclusion Criteria:

1. Be a PAYA-CS, defined as ≤39 years of age at the time of cancer diagnosis;
2. Be 18-45 years of age at the time of enrolment;
3. Received cancer treatment(s) with known cardiovascular risks (e.g., anthracyclines, trastuzumab, radiotherapy, platinum-based agents, vascular endothelial growth factor inhibitors, tyrosine kinase inhibitors);
4. Be cancer-free at the time of enrollment;
5. Stage B Heart Failure (SBHF)

   * In patients with availability of pre-treatment imaging:

     * ≥10% decrease in LVEF at post-treatment compared to pre-treatment
     * ≥15% decrease in GLS at post-treatment compared to pre-treatment
   * No pre-treatment imaging:

     * LVEF ≤53% in women/51% in men
     * GLS >-18%
     * Left ventricular hypertrophy (LV mass/body surface area: >95 g/m2 for women or >115 g/m2 for men)
     * Concentric remodelling (>0.42 relative wall thickness)
     * Diastolic dysfunction (≥ grade 1)
     * BNP ≥35pg/ml or NT-proBNP ≥125pg/ml

Exclusion Criteria:

1. Have an absolute or unresolved relative contraindication to exercise according to the American College of Sports Medicine guidelines;
2. Have an untreated physical or mental health concern that precludes safe and effective exercise participation;
3. Have established CVD (excluding mildly reduced LVEF as described above);
4. Be pregnant at time of recruitment;
5. Be currently engaging in frequent high-intensity exercise (>1 high-intensity exercise session per week);
6. Have substantial barriers to participating, including (1) living too far from study centre or (2) being unable or willing to comply with the study protocol.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 336 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Cardiorespiratory fitness | Baseline to 6-month follow-up (Primary RCT)
  Assessed via cardiopulmonary exercise test and quantified as VO2peak

SECONDARY OUTCOMES:
Cardiorespiratory fitness | Baseline to 24-month follow-up (Primary and Secondary RCTs)
  Assessed via cardiopulmonary exercise test and quantified as VO2peak
Ventilatory threshold | Baseline to 6-month follow-up (Primary RCT)
  Estimated using the V-slope method and according to the following criteria: i) an exaggerated response in the volume of carbon-dioxide (i.e., VCO2) relative to the volume of oxygen (i.e., VO2), and ii) the first identifiable break-point in in the minute ventilation (i.e., VE/VO2 vs work rate relationship).
Ventilatory threshold | Baseline to 24-month follow-up (Primary and Secondary RCTs)
  Estimated using the V-slope method and according to the following criteria: i) an exaggerated response in the volume of carbon-dioxide (i.e., VCO2) relative to the volume of oxygen (i.e., VO2), and ii) the first identifiable break-point in in the minute ventilation (i.e., VE/VO2 vs work rate relationship).
Anaerobic threshold | Baseline to 6-month follow-up (Primary RCT)
  Estimated according to the three-criterion discrimination technique: i) an excess VCO2 response relative to the VO2 response identified per the modified V-slope criteria; ii) the VE/VO2 to VO2 relationship having been flat or decreasing begins to increase without returning to baseline; and iii) there is no reciprocal decrease in PETCO2 at the point where PETO2 starts to rise systematically.
Anaerobic threshold | Baseline to 24-month follow-up (Primary and Secondary RCTs)
  Estimated according to the three-criterion discrimination technique: i) an excess VCO2 response relative to the VO2 response identified per the modified V-slope criteria; ii) the VE/VO2 to VO2 relationship having been flat or decreasing begins to increase without returning to baseline; and iii) there is no reciprocal decrease in PETCO2 at the point where PETO2 starts to rise systematically.
Post-exercise heart rate recovery | Baseline to 6-month follow-up (Primary RCT)
  One-minute HR recovery (HRR; an index of post-exercise parasympathetic reactivation) will be calculated as the HR-difference between peak exercise and following one minute of quiet standing on the treadmill immediately post-test.
Post-exercise heart rate recovery | Baseline to 24-month follow-up (Primary and Secondary RCTs)
  One-minute HR recovery (HRR; an index of post-exercise parasympathetic reactivation) will be calculated as the HR-difference between peak exercise and following one minute of quiet standing on the treadmill immediately post-test.
Left ventricular ejection fraction (LVEF) | Baseline to 6-month follow-up (Primary RCT)
  Assessed via 2D and 3D echocardiography
Left ventricular ejection fraction (LVEF) | Baseline to 24-month follow-up (Primary and Secondary RCTs)
  Assessed via 2D and 3D echocardiography
Global longitudinal strain (GLS) | Baseline to 6-month follow-up (Primary RCT)
  Assessed via 2D echocardiography
Global longitudinal strain (GLS) | Baseline to 24-month follow-up (Primary and Secondary RCTs)
  Assessed via 2D echocardiography
Early (E) and late (A) diastolic mitral inflow velocities and deceleration time | Baseline to 6-month follow-up (Primary RCT)
  Assessed via echocardiography
Early (E) and late (A) diastolic mitral inflow velocities and deceleration time | Baseline to 24-month follow-up (Primary and Secondary RCTs)
  Assessed via echocardiography
Early diastolic mitral septal and lateral annular velocities (e') | Baseline to 6-month follow-up (Primary RCT)
  Assessed via tissue Doppler imaging (TDI)
Early diastolic mitral septal and lateral annular velocities (e') | Baseline to 24-month follow-up (Primary and Secondary RCTs)
  Assessed via tissue Doppler imaging (TDI)
TR velocity | Baseline to 6-month follow-up (Primary RCT)
  Assess via spectral Doppler
TR velocity | Baseline to 24-month follow-up (Primary and Secondary RCTs)
  Assess via spectral Doppler
Left atrial volume | Baseline to 6-month follow-up (Primary RCT)
  Assess via 2D echocardiography
Left atrial volume | Baseline to 24-month follow-up (Primary and Secondary RCTs)
  Assess via 2D echocardiography
Diastolic function - E/e' ratio | Baseline to 6-month follow-up (Primary RCT)
  Calculated using the average of the TDI septal and lateral annular velocities (e')
Diastolic function - E/e' ratio | Baseline to 24-month follow-up (Primary and Secondary RCTs)
  Calculated using the average of the TDI septal and lateral annular velocities (e')
Left ventricular hypertrophy | Baseline to 6-month follow-up (Primary RCT)
  Assessed via Devereux formula and quantified as LV mass/body surface area: >95 g/m2 for women or >115 g/m2 for men
Left ventricular hypertrophy | Baseline to 24-month follow-up (Primary and Secondary RCTs)
  Assessed via Devereux formula and quantified as LV mass/body surface area: >95 g/m2 for women or >115 g/m2 for men
Concentric cardiac remodeling | Baseline to 6-month follow-up (Primary RCT)
  Assessed as >0.42 relative wall thickness
Concentric cardiac remodeling | Baseline to 24-month follow-up (Primary and Secondary RCTs)
  Assessed as >0.42 relative wall thickness
Resting heart rate | Baseline to 6-month follow-up (Primary RCT)
  Measured with an average of 2 readings taken via ECG during the resting period during the cardiac screening procedures.
Resting heart rate | Baseline to 24-month follow-up (Primary and Secondary RCTs)
  Measured with an average of 2 readings taken via ECG during the resting period during the cardiac screening procedures.
Resting systolic and diastolic blood pressure | Baseline to 6-month follow-up (Primary RCT)
  Calculated as average of 3 readings measured via automated sphygmomanometer per the Hypertension Canada guidelines.
Resting systolic and diastolic blood pressure | Baseline to 24-month follow-up (Primary and Secondary RCTs)
  Calculated as average of 3 readings measured via automated sphygmomanometer per the Hypertension Canada guidelines.
Apolipoprotein B | Baseline to 6-month follow-up (Primary RCT)
  Assessed via blood serum sample
Apolipoprotein B | Baseline to 24-month follow-up (Primary and Secondary RCTs)
  Assessed via blood serum sample
Total cholesterol | Baseline to 6-month follow-up (Primary RCT)
  Assessed via blood serum sample
Total cholesterol | Baseline to 24-month follow-up (Primary and Secondary RCTs)
  Assessed via blood serum sample
Low density lipoprotein | Baseline to 6-month follow-up (Primary RCT)
  Assessed via blood serum sample
Low density lipoprotein | Baseline to 24-month follow-up (Primary and Secondary RCTs)
  Assessed via blood serum sample
High density lipoprotein | Baseline to 6-month follow-up (Primary RCT)
  Assessed via blood serum sample
High density lipoprotein | Baseline to 24-month follow-up (Primary and Secondary RCTs)
  Assessed via blood serum sample
Whole body insulin sensitivity | Baseline to 6-month follow-up (Primary RCT)
  Assessed via Matsuda index
Whole body insulin sensitivity | Baseline to 24-month follow-up (Primary and Secondary RCTs)
  Assessed via Matsuda index
Hepatic insulin sensitivity | Baseline to 6-month follow-up (Primary RCT)
  Assessed via homeostasis model assessment insulin resistance (HOMA-IR)
Hepatic insulin sensitivity | Baseline to 24-month follow-up (Primary and Secondary RCTs)
  Assessed via homeostasis model assessment insulin resistance (HOMA-IR)
Pancreatic beta-cell function | Baseline to 6-month follow-up (Primary RCT)
  Assessed via the insulin secretion-sensitivity index-2 (ISSI-2)
Pancreatic beta-cell function | Baseline to 24-month follow-up (Primary and Secondary RCTs)
  Assessed via the insulin secretion-sensitivity index-2 (ISSI-2)
Body mass index | Baseline to 6-month follow-up (Primary RCT)
  Calculated as body weight (kg) divided by height (m) squared
Body mass index | Baseline to 24-month follow-up (Primary and Secondary RCTs)
  Calculated as body weight (kg) divided by height (m) squared
Objective physical activity | Baseline to 24-month follow-up (Primary and Secondary RCTs)
  Objectively assessed via wrist-worn physical activity/heart rate monitor to measure the intensity and duration of all planned and unplanned exercise during the study period
Subjective physical activity | Baseline to 6-month follow-up (Primary RCT)
  Subjectively assessed via Godin Leisure Time Physical Activity Questionnaire and reported as moderate-to-vigorous intensity physical activity (MVPA)
Subjective physical activity | Baseline to 24-month follow-up (Primary and Secondary RCTs)
  Subjectively assessed via Godin Leisure Time Physical Activity Questionnaire and reported as moderate-to-vigorous intensity physical activity (MVPA)
Social support | Baseline to 6-month follow-up (Primary RCT)
  Measured using the Social Support Survey-Clinical (SSS-C) form, a 5-item survey designed to measure five dimensions of social support + a single item to assess cancer-specific social support.
Social support | Baseline to 24-month follow-up (Primary and Secondary RCTs)
  Measured using the Social Support Survey-Clinical (SSS-C) form, a 5-item survey designed to measure five dimensions of social support + a single item to assess cancer-specific social support.
Exercise self-efficacy | Baseline to 6-month follow-up (Primary RCT)
  Measured using the Multidimensional Self-Efficacy for Exercise Scale (MSES) to measure three behavioural subdomains: task, scheduling, and coping
Exercise self-efficacy | Baseline to 24-month follow-up (Primary and Secondary RCTs)
  Measured using the Multidimensional Self-Efficacy for Exercise Scale (MSES) to measure three behavioural subdomains: task, scheduling, and coping
Anxiety | Baseline to 6-month follow-up (Primary RCT)
  Measured using the Generalized Anxiety Disorder (GAD-7), a 7-item inventory that assesses 2-week anxiety symptom frequency on a 0-3 scale, with higher scores reflecting higher symptom frequency. A cut-off of ≥10 indicates some degree of clinical anxiety.
Anxiety | Baseline to 24-month follow-up (Primary and Secondary RCTs)
  Measured using the Generalized Anxiety Disorder (GAD-7), a 7-item inventory that assesses 2-week anxiety symptom frequency on a 0-3 scale, with higher scores reflecting higher symptom frequency. A cut-off of ≥10 indicates some degree of clinical anxiety.
Depression | Baseline to 6-month follow-up (Primary RCT)
  Measured using the Patient Health Questionnaire (PHQ-9), a 9-item inventory that assesses 2-week depressive symptom frequency on a 0-3 scale, with higher scores reflecting higher symptom frequency. The PHQ-9 has been validated in cancer survivors using a cut-off of ≥8 to indicate some degree of clinical depression.
Depression | Baseline to 24-month follow-up (Primary and Secondary RCTs)
  Measured using the Patient Health Questionnaire (PHQ-9), a 9-item inventory that assesses 2-week depressive symptom frequency on a 0-3 scale, with higher scores reflecting higher symptom frequency. The PHQ-9 has been validated in cancer survivors using a cut-off of ≥8 to indicate some degree of clinical depression.
Health-related quality of life | Baseline to 6-month follow-up (Primary RCT)
  Measured using the Medical Outcomes Survey Short-Form (SF-12).
Health-related quality of life | Baseline to 24-month follow-up (Primary and Secondary RCTs)
  Measured using the Medical Outcomes Survey Short-Form (SF-12).
Health service utilization | Baseline to 6-month follow-up (Primary RCT)
  Measured using the Health Service Utilization Inventory.
Health service utilization | Baseline to 24-month follow-up (Primary and Secondary RCTs)
  Measured using the Health Service Utilization Inventory.

OTHER OUTCOMES:
Therapeutic alliance | Baseline to 6-month follow-up (Primary RCT)
  Measured using the Working Alliance Inventory Short-Revised (WAI-SR) form.
Testing Performance | Study initiation to end of 66-month study period (Primary and Secondary RCTs)
  Defined as the percent of tests that achieve 'peak' termination criteria relative to the total number of tests completed across all time points
Serious and non-serious adverse events | Study initiation to end of 66-month study period (Primary and Secondary RCTs)
  Defined as the number and frequency of testing-, intervention-, and non-intervention-related serious (i.e. Grade 3 to 5; NCI-CTCAE criteria) and non-serious (i.e. Grade 1 to 2; NCI-CTCAE criteria)
Exercise Adherence | Study initiation to end of 48-month phase I intervention period (Primary RCT - CORE participants)
  This variable applies only to CORE participants. Exercise adherence is defined as the relative dose intensity (i.e. the percent of total dose of exercise performed, relative to the total dose prescribed) and quantified according to metabolic equivalents.
Medication Compliance | Study initiation to end of 48-month phase I intervention period (Primary RCT - CORE participants)
  Defined as the percent of pharmaceutical doses taken based on the total number of doses prescribed (applicable only to those that are provided pharmaceutical therapy for CVD risk factor modification)
Behavioural Compliance | Study initiation to end of 66-month study period (Primary RCTs - CORE participants)
  Defined as the percent of behavioural support resources accessed, based on the number recommended (one per month)
Oxygen utilization during HIIT | Study initiation to end of 48-month phase I intervention period (CORE substudy participants; Primary RCT)
  Quantified as timepoint measures of oxygen utilization assessed via portable metabolic measurement system within the final 30 seconds of the warm-up, work and recovery periods, and the cool down during pre-specified high-intensity interval training sessions
Power output during HIIT | Study initiation to end of 48-month phase I intervention period (CORE sub-study participants; Primary RCT)
  Quantified as power output (watts) assessed cycle ergometer within the final 30 seconds of the warm-up, work and recovery periods, and the cool down during pre-specified high-intensity interval training sessions
Heart rate response during HIIT | Study initiation to end of 48-month phase I intervention period (CORE sub-study participants; Primary RCT)
  Quantified via heart rate monitor or single-lead ECG within the final 30 seconds of the warm-up, work and recovery periods, and the cool down during pre-specified high-intensity interval training sessions
Energy expenditure during HIIT | Study initiation to end of 48-month phase I intervention period (CORE sub-study participants; Primary RCT)
  Quantified as total metabolic equivalent of task following HIIT sessions
Perceived exertion during HIIT | Study initiation to end of 48-month phase I intervention period (CORE sub-study participants; Primary RCT)
  Assessed via rating of perceived exertion scale (6-20) within the final 30 seconds of the warm-up, work and recovery periods, and the cool down during pre-specified high-intensity interval training sessions
Felt arousal during HIIT | Study initiation to end of 48-month phase I intervention period (CORE sub-study participants; Primary RCT)
  Affective arousal is evaluated via the felt arousal scale that assesses energy/arousal level on a scale of 1 (low arousal) to 6 (high arousal) within the final 30 seconds of the warm-up, work and recovery periods, and the cool down during pre-specified HIIT sessions
Feeling affect during HIIT | Study initiation to end of 48-month phase I intervention period (CORE sub-study participants; Primary RCT)
  The feeling scale is used to assess affective valence (pleasure/displeasure; feeling good/bad) on a scale of -5 (vey bad) to +5 (very good) within the final 30 seconds of the warm-up, work and recovery periods, and the cool down during pre-specified high-intensity interval training sessions
Resilience | Study initiation to end of 48-month phase I intervention period (CORE sub-study participants; Primary RCT)
  Measured using the Brief Relilience Scale (BRS), a 6-item inventory that assesses recovery, resistance, adaptation, and thriving.
Stress | Study initiation to end of 48-month phase I intervention period (CORE sub-study participants; Primary RCT)
  Measured using two items based on the Canadian Community Health Survey assessing the average daily stress experienced that day and over the past week.
Feeling states | Study initiation to end of 48-month phase I intervention period (CORE sub-study participants; Primary RCT)
  Assessed via ecological momentary assessments using brief reports completed 6 times a day on intervention weeks 1, 7, 16, 22, four weeks post intervention, and 26 weeks post intervention

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Toronto, Ontario, Canada